CLINICAL TRIAL: NCT04235335
Title: Healing Circles: An Evaluation of an Intervention for Canadian Indigenous Mothers and Children Affected by Intimate Partner Violence
Brief Title: Healing Circles: An Intervention for Canadian Indigenous Mothers & Children Affected by IPV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Caroline Piotrowski, Associate Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2019:501
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Violence, Domestic
Keywords: domestic violence; exposure to violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wait List Control (Other): Participants receive intervention after 12 week delay
  Interventions: Behavioral: Indigenous Mother's Empowerment Program & Indigenous Kid's Club Program

INTERVENTIONS:
Behavioral: Indigenous Mother's Empowerment Program & Indigenous Kid's Club Program — Weekly groups administered to mothers and children simultaneously but separately for 10 weeks

SUMMARY:
Evaluation of Mother's Empowerment Program and Kid's Club Program adapted specifically for Indigenous mothers and children affected by intimate partner violence in Canada

DETAILED DESCRIPTION:
Research Goals & Objectives. Our overall goal is to conduct a feasibility study of two successful evidence-based interventions (Mother's Empowerment Program and Kid's Club Program) designed specifically to meet the needs of Indigenous mothers and their children who have experienced intimate partner violence (IPV).

Specifically, our objectives are:

1. To successfully adapt two existing effective evidence-based interventions for mothers and children who have experienced IPV for Indigenous mothers and children who have experienced IPV. Our adaptation process reflects our overall integrated knowledge translation (iKT) approach, undertaken in close partnership with our Community Advisory Council (CAC) and in consultation with Elders at both sites. As outlined by the Canadian Institutes of Health Research (CIHR), it follows a two-eyed seeing approach, incorporating Western and Indigenous knowledge, ways of knowing and being.
2. To pilot and evaluate our adapted interventions with mothers and children recruited from our community partners (Wahbung Abinoonjiiag, an Indigenous non-profit organization in Winnipeg and Discovery House, a crisis shelter and second stage housing facility for women in Calgary). We plan to evaluate our adapted programs using a two-eyed seeing approach that combines Western (quantitative) and Indigenous (qualitative) methodologies. As part of our iKT approach, our mixed methods evaluation will rely upon ongoing engagement and feedback from our CAC. Quantitative methods (e.g., standardized questionnaires) will be used to assess changes in the mental and physical health and well-being of mothers and their children over time. Qualitative methods (e.g., semi-structured interviews, narratives) will be used to evaluate the intervention experience and perceived changes in self perceptions (e.g., resilience).

Hypotheses. We will determine if there is an increase, both immediately post-intervention and sustained over 6-8 months, in mothers' and children's mental (e.g., resilience) and physical well-being (e.g., perceived health status), and if there is a reduction in mothers' and children's mental health (e.g., depression, anxiety and traumatic stress symptoms) and physical difficulties (e.g., somatic symptoms such as headaches). For children, analyses will take age, gender and sex into account.

ELIGIBILITY:
Inclusion Criteria:

* mothers self-reported experience of past intimate partner violence, English-speaking, with at least one school-aged child

Exclusion Criteria:

-

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Maternal Depression | Measured immediately post-intervention
  Centers for Epidemiological Studies-Depression (CES-D)
Maternal Depression | Measured 6-8 months post-intervention
  Centers for Epidemiological Studies-Depression (CES-D)
Child Depression | Measured Immediately post-intervention
  Child Depression Inventory (CDI)
Child Depression | Measured 6-8 months post-intervention
  Child Depression Inventory (CDI)
Maternal Anxiety | Measured Immediately post-intervention
  Beck Anxiety Scale
Maternal Anxiety | Measured 6-8 months post-intervention
  Beck Anxiety Scale
Child Anxiety | Measured immediately post-intervention
  Revised Children's Manifest Anxiety Scale - 2nd Edition Short Form (RCMAS-2)
Child Anxiety | Measured 6-8 months post-intervention
  Revised Children's Manifest Anxiety Scale - 2nd Edition Short Form (RCMAS-2)
Maternal trauma symptoms | Measured immediately post-intervention
  PTSD Checklist (PCL-5)
Maternal trauma symptoms | Measured 6-8 months post-intervention
  PTSD Checklist (PCL-5)
Child trauma symptoms | Measured immediately post-intervention
  University of California - Los Angeles (UCLA) Reaction Index
Child trauma symptoms | Measured 6-8 months post-intervention
  University of California - Los Angeles (UCLA) Reaction Index

SECONDARY OUTCOMES:
Maternal resilience | Measured immediately post-intervention
  Adult Resilience Measure - revised (ARM-R)
Maternal resilience | Measured 6-8 months post-intervention
  Adult Resilience Measure - revised (ARM-R)
Child resilience | Measured immediately post-intervention
  Child & Youth Resilience Measure - revised (CYRM-R)
Child resilience | Measured 6-8 months post-intervention
  Child & Youth Resilience Measure - revised (CYRM-R)
Maternal social support | Measured immediately post-intervention
  Inventory of Socially Supportive Behaviors
Maternal social support | Measured 6-8 months post-intervention
  Inventory of Socially Supportive Behaviors
Maternal self esteem | Measured immediately post-intervention
  Rosenberg Self Esteem Scale
Maternal self esteem | Measured 6-8 months post-intervention
  Rosenberg Self Esteem Scale

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Piotrowski, PhD MPH, Principal Investigator — University of Manitoba
Locations (1):
- Discovery House, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Graham-Bermann SA, Miller-Graff L. Community-based intervention for women exposed to intimate partner violence: A randomized control trial. J Fam Psychol. 2015 Aug;29(4):537-47. doi: 10.1037/fam0000091. PMID 26030027
- [Result] Graham-Bermann SA, Miller-Graff LE, Howell KH, Grogan-Kaylor A. An Efficacy Trial of an Intervention Program for Children Exposed to Intimate Partner Violence. Child Psychiatry Hum Dev. 2015 Dec;46(6):928-39. doi: 10.1007/s10578-015-0532-4. PMID 25596929
- [Result] Graham-Bermann SA, Lynch S, Banyard V, DeVoe ER, Halabu H. Community-based intervention for children exposed to intimate partner violence: an efficacy trial. J Consult Clin Psychol. 2007 Apr;75(2):199-209. doi: 10.1037/0022-006X.75.2.199. PMID 17469878